CLINICAL TRIAL: NCT04086771
Title: Southeast Asian Women's Health Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of South Florida (Other); American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Jennifer Kue, Associate Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018B0521
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Cervical Cancer
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Intervention group- Tailored Navigation Delivered by Community Health Advisor (CHA+TN)
  Control Group- Information and Reminder Only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Navigation) (Experimental): Participants will be contacted by CHAs by phone one week after giving informed consent and completion of the baseline survey. CHAs will contact participants once a week for up to 10 weeks (a maximum of 10 attempts or until a clinic appointment is made, whichever comes first). Using the TIMS© message library, the CHAs will engage participants in conversations about breast and cervical cancer screening and navigate the participants to overcome any barriers to screening and motivate them to make a clinic appointment. Personal messages from mothers to daughters and vice versa and screening reminder notecards will be sent at 12-months (T3). At 18-months (T4), CHAs will follow-up with navigation group participants who reported completing a mammogram during the navigation process. Screening completion will be measured by self-report and confirmed via medical record check.
  Interventions: Behavioral: Navigation
- Control Group (Information only) (Placebo Comparator): Participants will be mailed an informational brochure on mammography and Pap testing one week after enrollment into the study. At 3-months post enrollment, CHAs will conduct a follow-up phone call with each participant to assess mammogram and/or Pap testing completion (primary outcomes). At 12-months (T3) post enrollment, CHAs will contact all control group participants by phone to confirm a scheduled appointment or screening completion. For those who completed a mammogram within the 12 months since enrollment, generic screening reminder notecards will be sent by mail. At 18-months (T4), CHAs will follow-up with those control group participants who reported scheduling a mammogram, Pap smear, or both at the 12-month (T3) time point.
  Interventions: Other: Information only

INTERVENTIONS:
Behavioral: Navigation — Weekly phone-calls, personal messages, and American Cancer Society Pap test and mammography test reminder post card
  Arms: Intervention Group (Navigation)
Other: Information only — American Cancer Society breast and cervical cancer screening information and Pap test and mammography test reminder post card
  Arms: Control Group (Information only)

SUMMARY:
Cancer is the leading cause of death for Southeast Asian refugee and immigrant (R/I) women; yet they have unacceptably low screening rates. Drawing on successful tailored navigation interventions, the purpose of this study is to compare a culturally congruent, tailored navigation intervention delivered by bilingual and bicultural Community Health Advisors (CHAs) to increase age-appropriate breast and cervical cancer screening completion among intergenerational Southeast Asian R/I women (mother-daughter dyads) with information and reminder only. We will examine the underlying factors that associate with the intervention that influence cancer screening completion. We will also explore the influence of intergenerational exchange of breast and cervical cancer screening information between mothers and daughters. This multi-faceted intervention, combining culturally tailored messages and navigation via CHAs, has high potential for scalability across settings and diseases for hard-to-reach populations. In addition, this study focuses on breast and cervical cancer screening jointly potentially increasing the public health impact.

DETAILED DESCRIPTION:
Cancer is the leading cause of death for Southeast Asian refugee and immigrant women. Cambodian, Lao, and Vietnamese (hereafter referred to as SEAR/I) women have disproportionately high incidence rates of breast and cervical cancers. Breast cancer incidence increased significantly for all Asians from 1988 to 2013, but the largest increase was in SEAR/I women (APC=2.5, 95% CI 0.8, 4.2). Over the past two decades, SEAR/I women experienced significant increases in breast cancer incidence across age groups compared to other Asian and White women. Lao and Cambodian women are 2.5 times and Vietnamese women are 40% more likely to be diagnosed with cervical cancer than are White women. Despite evidence that regular screening through mammography and Pap testing reduces breast and cervical cancer mortality, SEAR/I women continue to have strikingly low rates of screening (75.4% for Pap tests and 64.1% for mammography), well below the Healthy People 2020 target of 93% and 81.1%, respectively. Drawing on successful tailored navigation interventions, the purpose of this study is to test the efficacy of a culturally-relevant, tailored navigation intervention delivered through bilingual and bicultural Community Health Advisors (CHAs) for intergenerational SEAR/I women (mother-daughter dyads). Ethnically matched CHAs will use the tested Tailored Intervention Messaging System (TIMS©) to educate and navigate participants from the community to health clinic to complete mammography and/or Pap testing.

Our specific aims are to:

AIM 1: Test the efficacy of tailored navigation intervention delivered by SEA community health advisors (CHA+TN) to increase age-appropriate breast and cervical cancer screening completion compared to an information and reminder only control among intergenerational SEAR/I dyads.

H1: The intervention group (CHA+TN) will have significantly higher age-appropriate breast and cervical cancer screening rates compared with the control group (information + reminder only).

AIM 2: Examine the underlying mechanisms (both mediating and moderating factors) associated with the intervention (CHA+TN) that influence breast and cervical cancer screening completion.

Exploratory AIM 3: Explore in greater detail the influence of intergenerational exchange of information between mothers and daughters related to breast and cervical cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* Live in Ohio
* Self-identify as Filipino, Cambodian, Lao, or Vietnamese
* Aged 21 years and older
* Non-adherent for mammogram, Pap test, or both
* Have a mother or daughter aged 21 years and older.
* If potential participants do not have a mother or daughter, then they would have to have an immediate female family member, such as an aunt, niece, or grandmother aged 21 years and older who could also be recruited into the study.

Exclusion Criteria:

* Women who have been previously diagnosed with breast and/or cervical cancer.
* Siblings such as a sister will not be considered eligible unless they are from different generations.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Mammogram test completion | 18 months
  Screening completion measured by self-report
Pap test completion | 18months
  Screening completion measured by self-report

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kue, PhD, Principal Investigator — University of South Florida; Judith Tate, PhD, RN, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No